CLINICAL TRIAL: NCT03427372
Title: The Effect of Anxiety and Depression Mood on Post Spinal Puncture Headache and Backache
Brief Title: The Effect of Psychological State on Post Spinal Puncture Headache and Backache
Status: Completed | Type: Observational
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Kevser Peker, MD, Ahi Evran University Education and Research Hospital
Other Study IDs: post dural puncture headache
Record Dates: First submitted 2018-02-03; First posted 2018-02-09 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1: patients with headache: the patients who have post spinal puncture headache after spinal anesthesia
  Interventions: Behavioral: anxiety scale, depression scale
- group 2: patients without headache: the patients who do not have post spinal puncture headache after spinal anesthesia
  Interventions: Behavioral: anxiety scale, depression scale
- group 3: patients with backache: the patients who have post spinal puncture backache after spinal anesthesia
- group 4: patients without backache: the patients who do not have post spinal puncture backache after spinal anesthesia

INTERVENTIONS:
Behavioral: anxiety scale, depression scale — post spinal puncture headache and backache will be assess by using visual analogue scale, anxiety will assess by beck anxiety scale, depression mood will assess by beck depression scale
  Groups: group 1: patients with headache; group 2: patients without headache

SUMMARY:
To investigate the effect of patient mood before spinal anesthesia on post spinal puncture headache and backache

DETAILED DESCRIPTION:
Before spinal anesthesia patients' anxiety and depression mood will recorded with Beck anxiety and Beck depression scale fifteen minute before spinal anesthesia.Seven days after surgery post spinal puncture headache and backache will assess by a telephonic interview

ELIGIBILITY:
Inclusion Criteria:

* patient scehedule surgery under spinal anesthesia
* between 18-80 years old

Exclusion Criteria:

* patients with psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-80 years old American Society of Anesthesiology (ASA) I-III patients underwent spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
post spinal puncture headache (PDPH) | one week after surgery
  For assessing PDPH, patients will ask whether they experienced headache through the use of a dichotomous scale (yes or no answer). The severity of PDPH will be assessed by the Dittmann's scale. This PDPH specific scale was composed of 4 levels of severity. Level 1 indicated minimal PDPH with no use of medications to manage PDPH with the patient able to participate in daily living activities without any inferences. Level 2 indicated mild PDPH that required the use of analgesics with patients still able to engage in daily living activities. Level 3 indicated moderate PDPH where analgesic administration was required to control the level of pain. Level 4 indicated severe PDPH with an epidural blood patch recommended.

SECONDARY OUTCOMES:
anxiety | fifteen minutes before spinal anesthesia
  Anxiety will evaluated by the Beck Anxiety Inventory (BAI), which consists of 21 questions about how the individual has felt in the preceding week regarding common anxiety symptoms, such as sweating, tremor, fear, and feelings of distress. The cutoff point for anxiety is 12, and scores between 1 and 11 are considered subsyndromal anxiety.
depression | fifteen minutes before spinal anesthesia
  Depression will assess by beck depression scale. The Beck Depression Scale (BDS) uses a 3-point Likert type response scale to 21 questions. In the scale, a total of 0-13 points are considered 'normal', 14-25 points to indicate 'depression', and 26-63 points to indicate'severe depression'.
post spinal puncture backache (PDPB) | one week after surgery
  The presence of backache will asses by using visual analogue scale (VAS). Patients will familiarized with 10 cm marked VAS for assessment of back pain, where 0 cm defines no pain, and 10 cm defines the maximum intolerable pain

CONTACTS AND LOCATIONS:
Overall Officials: kevser peker, Principal Investigator — Ahi Evran University Education and Research Hospital
Locations (1):
- Ahi evran university education and research hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peker K, Polat R. The effects of preoperative reactions of emotional distress on headache and acute low back pain after spinal anesthesia: A prospective study. J Psychosom Res. 2021 May;144:110416. doi: 10.1016/j.jpsychores.2021.110416. Epub 2021 Mar 11. PMID 33735647